CLINICAL TRIAL: NCT00532857
Title: Phase II Study of Primary Chemotherapy With Paclitaxel, Gemcitabine, and Trastuzumab in Patients With HER2 Positive Operable Breast Cancer
Brief Title: Phase II Study of Primary Chemotherapy With Paclitaxel, Gemcitabine, and Trastuzumab
Acronym: PGH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jungsil Ro (Other Government)
Responsible Party: Sponsor-Investigator, Jungsil Ro, Chief, Center for Clinical Trials, National Cancer Center, Korea, National Cancer Center, Korea
Organization: National Cancer Center, Korea (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-06-235
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2012-01-04 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
Keywords: Patients with HER2 + stage II/III breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Gemcitabine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel/Gemcitabine/Trastuzumab (Experimental)
  Interventions: Drug: Paclitaxel/Gemcitabine/Trastuzumab

INTERVENTIONS:
Drug: Paclitaxel/Gemcitabine/Trastuzumab — 80 mg/m2 of paclitaxel 1,200 mg/m2 of gemcitabine, day 1, day 8 every 3-week. trastuzumab at a dose of 4 mg/kg IV on D1 of first treatment cycle subsequently given weekly at a dose of 2 mg/kg
  Other Names: Paclitaxel; Gemzar; Herceptin

SUMMARY:
To evaluate the pathologic complete response rate to preoperative administration of Paclitaxel, Gemcitabine, and Trastuzumab (HerceptinÒ) (PGH)

DETAILED DESCRIPTION:
Primary objectives: To evaluate the pathologic complete response rate to preoperative administration of Paclitaxel, Gemcitabine, and Trastuzumab (HerceptinÒ) (PGH) Secondary objectives: To assess breast conserving rate after preoperative chemotherapyTo evaluate clinical response rate, disease free survival (DFS), and overall survival (OS) To assess the safety profiles of PGH

Treatment will be delivered in the outpatient setting. Each three-week cycle consists of paclitaxel 80 mg/m2 (day 1, 8) and gemcitabine 1200 mg/m2 (day1, 8) in addition to trastuzumab, which is given at a dose of 4 mg/kg IV on day 1 of the first treatment cycle over 90 min, and subsequently given weekly at a dose of 2 mg/kg over 30 min. Patients will receive 6 cycles of therapy unless there is any evidence of no response suitable for operation(SD or PD) or unacceptable toxicity or noncompliance by patient with protocol requirements. Patients who are unsuitable for op due to SD or PD, will undergo XRT. However, when patients are still suitable for op even with SD or PD, these patients will undergo op.Such decision will be made at physician's discretion at each institution. Also, even though there is neither clear evidence of disease progression nor severe toxicity, if patient declines the treatment, study treatment can be discontinued. Response will be documented by physical examination, sonography and/or chest CT prior to treatment and every three cycles. Postoperatively within 1-3 week, trastuzumab 6 mg/kg every 3 weeks x 11 and tamoxifen or AI for 5 years will be given as indicated. Radiation therapy will be initiated postoperatively in 3-4 weeks according to the standard practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically confirmed and newly diagnosed operable breast cancer
* HER2 positive (all FISH +)
* Axillary node positive (by PET or cytologically determine node by sonography) and/or tumor size > 5 cm -No prior hormonal, chemotherapy or radiotherapy is allowed.
* No breast operation other than biopsy to make diagnosis is allowed.
* Age: 18-years and older, not pregnant pre-, and postmenopausal women with good performance status (ECOG 0-1)
* Adequate hematopoietic function:

Absolute granulocyte count ³1500/mm3,

* platelet ³100,000/mm3, Hemoglobin ³ 10 g/mm3
* Adequate renal function: Serum creatinine £ 1.5 mg/dl
* Adequate hepatic function: total bilirubin: £ 1.5 mg/dl, AST/ALT: £ 2 times normal, Alkaline phosphatase: £ 2 times normal-Adequate cardiac function:

  1. normal or nonspecific EKG taken within 1 mo of enrollment
  2. LVEF ³ 50% by MUGA or Echocardiogram taken within 1 mo of enrollment
* Normal mental function to understand and sign the consent

Exclusion Criteria:

* patients who received hormonal, chemotherapy or radiotherapy for breast cancer
* patients who underwent surgery for breast cancer
* patients with a history of uncompensated congestive heart failure
* Patients with node-negative stage IIA (T2N0) breast cancer
* Patients who have history of cancer other than in situ uterine cervix cancer or nonmelanotic skin cancer

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-03; Primary Completion 2008-02 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the pathologic complete response rate To assess breast conserving rate after preoperative chemotherapy To evaluate clinical response rate, disease free survival (DFS), and overall survival (OS) To assess the safety profiles of PGH | Prospective: a protocol that observes events in real time (may occur in the future)

CONTACTS AND LOCATIONS:
Overall Officials: Jungsil Ro, MD,PhD, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, 809 Madu1-dong, Ilsandong-gu, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Im SA, Lee KS, Ro J, Lee ES, Kwon Y, Ahn JH, Ahn JS, Kim JH, Kang HS, Shin KH, Noh DY, Park IA, Kim SB, Im YH, Ha SW. Phase II trial of preoperative paclitaxel, gemcitabine, and trastuzumab combination therapy in HER2 positive stage II/III breast cancer: the Korean Cancer Study Group BR 07-01. Breast Cancer Res Treat. 2012 Apr;132(2):589-600. doi: 10.1007/s10549-011-1852-0. Epub 2011 Nov 18. PMID 22094934